CLINICAL TRIAL: NCT00314964
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Study Evaluating PD-0299685 for Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Study Evaluating PD-0299685 for the Treatment of Vasomotor Symptoms (Hot Flashes / Flushes) Associated With Menopause
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4291023
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: PD-0299685

SUMMARY:
The primary purpose of this study is to determine if PD-0299685 is effective and safe in the treatment of vasomotor symptoms (hot flashes / flushes) associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal as defined by 6 months of spontaneous amenorrhea with serum FSH levels >40mlU/ml and estradiol < than = 25 pg/mL or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy and FSH levels > 40 mlU/ml and estradiol < than = 25 pg/mL
* Women reporting at least 50 moderate to severe vasomotor symptoms per week, recorded for seven consecutive days
* Aged 40 to 70 years

Exclusion Criteria:

* No estrogen monotherapy or estrogen/progesterone containing drug products within applicable wash out period prior to screening
* Use of SERMs, clonidine within 4 weeks of screening
* Use of CNS active medication within 1 week of screening
* Use of medications (SSRI; SNRI), herbal or dietary supplements, including black cohosh, soy, phytoestrogens or over the counter agent known to possibly be effective for the treatment of vasomotor symptoms, within 4 weeks of screening
* Participation in clinical trial within 30 days
* Significant medical or psychiatric illness within past 12 months

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2006-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of PD-0299685 in reducing both the frequency and severity of vasomotor symptoms, from baseline to week 4 and week 12.

SECONDARY OUTCOMES:
To assess the safety profile of PD-0299685; the benefit of PD-0299685 in quality of life measures and treatment satisfaction of PD-0299685, when compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (68):
- United States (44):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Alanta, Georgia
  - Pfizer Investigational Site, Alpharetta, Georgia
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Stockbridge, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Waconia, Minnesota
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Springfeild, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Lawrenceville, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, New Bern, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
- Australia (4):
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Dulwich, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Subiaco, Western Australia
- Canada (5):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- France (4):
  - Pfizer Investigational Site, Montpellier, Cedex 5
  - Pfizer Investigational Site, Évry
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
- South Africa (7):
  - Pfizer Investigational Site, Central, Port Elizabeth, Eastern Cape
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Midrand, Gauteng
  - Pfizer Investigational Site, Radiokop, Gauteng
  - Pfizer Investigational Site, Dundee, KwaZulu-Natal
  - Pfizer Investigational Site, Westville, KwaZulu-Natal
  - Pfizer Investigational Site, Parow, Western Cape
- Spain (4):
  - Pfizer Investigational Site, Gavà, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Valencia, Valencia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4291023&StudyName=Study%20evaluating%20PD-0299685%20for%20the%20treatment%20of%20vasomotor%20symptoms%20%28Hot%20Flashes%20/%20Flushes%29%20associated%20with%20menopause